CLINICAL TRIAL: NCT00384631
Title: Intravitreal Bevacizumab for Neovascular Glaucoma; a Randomized Placebo Controlled Clinical Trial
Brief Title: Intravitreal Bevacizumab for Neovascular Glaucoma
Acronym: IVB NVG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8414
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Neovascular; Glaucoma
Keywords: Neovascular; Glaucoma; Bevacizumab; Avastin; Intravitreal; IOP
MeSH Terms: conditions — Glaucoma | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Sham Comparator)
  Interventions: Other: subconjunctival normal saline
- 1 (Experimental)
  Interventions: Drug: Avastin

INTERVENTIONS:
Other: subconjunctival normal saline — 0.1cc normal saline injection in the subconjunctival space repeated twice at monthly intervals
  Arms: 2
Drug: Avastin — intravitreal injection of avastin 2.5mg repeated twice at monthly intervals
  Arms: 1

SUMMARY:
Several studies have confirmed high levels of vascular endothelial growth factor (VEGF) in eyes with neovascular glaucoma (NVG). The role of VEGF inhibitors in regression of other neovascular disorders such as wet-type age-related macular degeneration and diabetic macular edema has been described. We aim to evaluate the effect of three intravitreal injections of bevacizumab (Avastin) 2.5 mg versus a sham procedure for treatment of NVG. Outcome measures include intraocular pressure and extent of iris neovascularization. Both study arms will receive conventional treatment for NVG.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NVG
* Vision less than 20/200
* age 10-80 years

Exclusion Criteria:

* Uncontrolled Blood Pressure
* History of thromboembolism
* Congestive Heart Failure
* Renal Failure
* Pregnancy or Lactation
* Active ocular or periocular infection
* No light perception

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-04; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in intraocular pressure | 6 months
Change in extent of iris neovascularization | 6 months

SECONDARY OUTCOMES:
Best corrected visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Yazdani, MD, Principal Investigator — Ophthalmic Research Center, Shaheed Beheshti Medical University
Locations (1):
- Labbafinejad Medical Center, Tehran, Tehran Province, Iran